CLINICAL TRIAL: NCT05344755
Title: Investigation of the Effect of Plantar Sensory Training on Pain, Foot Posture, Functional Activities, Gait and Balance Parameters in Individuals With Hallux Valgus
Brief Title: Effects of Plantar Sensory Training in Individuals With Hallux Valgus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Kırdı, Principal İnvestigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20014
Record Dates: First submitted 2022-03-26; First posted 2022-04-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hallux Valgus; Pain; Balance; Distorted
Keywords: hallux valgus; pain; sensory training; plantar sensory
MeSH Terms: conditions — Hallux Valgus; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plantar Sensorial Training (Experimental): In addition to hallux valgus mobilization, active thumb abduction, strengthening of the muscles around the feet, hallux valgus taping and hallux valgus night splint, sensory training (using deep plantar massage, brushing, dipping techniques) will be performed.
  Interventions: Other: Plantar Sensorial Training
- Control Group (Active Comparator): Routine hallux valgus physiotherapy approaches such as: hallux valgus mobilization, active thumb abduction, strengthening of the muscles around the feet, hallux valgus taping and hallux valgus night splint.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Plantar Sensorial Training — In addition to the routine treatment, plantar sensorial training will be added.
  Arms: Plantar Sensorial Training
Other: Control Group — Routine physiotherapy management of the Hallux valgus
  Arms: Control Group

SUMMARY:
Hallux valgus is a forefoot deformity with a high prevalence, which can progress to lateral deviation of the big toe, medial deviation of the first metatarsal, and subluxation of the first metatarsophalangeal joint in the future. It has been reported in studies that changes in the load distribution of the foot in hallux valgus patients, hyperkeratosis, especially first-line pain, and sensory receptors on the sole of the foot may result in the effect of sensory receptors on the sole of the foot, and thus the balance may be negatively affected, poor postural stability and an increase in the risk of falling. It is thought that increased sensitivity to the senses coming from the feet with sensory training can improve the balance and reduce the risk of falling as a result of better perception of foot orientation and position.

DETAILED DESCRIPTION:
Achieving balance depends on the visual, vestibular and somatosensory systems working together and in interaction. One of the important components of the somatosensory system is the cutaneous receptors. Merkel discs, Paccini corpuscles, Meissner corpuscles and Ruffini endings are located on the plantar surface of the foot, which makes contact with the ground. Plantar cutaneous receptors are sensitive to pressure during ground contact and provide site-specific information for cortical mapping and may affect postural responses. It is recommended that sensory training of the sole of the foot, rough insoles and transcutaneous electrical stimulation applications should be added to rehabilitation in order to increase the afferent sensory feedback from the sole of the foot in patients with multiple sclerosis, starting from the early stages of the disease. It has been reported in studies that the sensory input of different foot regions has an important role in the transition and timing of the stance and swing phase in gait. It has been suggested that cutaneous reflexes in the foot can provide functional locomotion and modulation of lower extremity flexor and extensor muscle activity. It has been reported in studies that changes in the load distribution of the foot in hallux valgus patients, hyperkeratosis, especially first-line pain, and sensory receptors on the sole of the foot may result in the effect of sensory receptors on the sole of the foot, and thus the balance may be negatively affected, poor postural stability and an increase in the risk of falling. It is thought that increased sensitivity to the senses coming from the feet with sensory training can improve the balance and reduce the risk of falling as a result of better perception of foot orientation and position. Therefore, the aim of our study; It was determined as the examination of the effect of plantar sensory training on pain, foot posture, functional activities, gait and balance parameters in individuals with hallux valgus.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mild or moderate hallux valgus;
* Volunteer to participate in the study

Exclusion Criteria:

* Having pathologies that may cause sensory problems such as diabetes, multiple sclerosis, myelomeningocele, severe disc herniation,
* Having an orthopedic, rheumatological or neurological disease other than hallux valgus that will prevent participation in the exercise program
* Having previous foot surgery,
* Having a cooperation problem at a level that cannot understand and apply the exercises.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Foot-Related pain assessment | change from baseline pain severity at 6 weeks
  Visual Analogue Scale will be used to evaluate the pain severity of individuals. Participants will be asked to mark their pain at rest and activity on a horizontal line of 100 millimeters, with 100 indicating maximum pain and 0 indicating no pain.

SECONDARY OUTCOMES:
Change in Light touch sensation | change from baseline light touch sensation at 6 weeks
  The light touch sense of the sole of the foot will be evaluated with the Semmes-Weinstein monofilament test. This test is widely used to evaluate light touch and pressure sense. The response to touch is tested with monofilaments of varying thickness and diameter, and the value that the patient feels is recorded.
Change in foot function | change from baseline foot function at 6 weeks
  The AOFAS Hallux-Metatarsophalangeal-Interphalangeal Scale created by the American Foot and Ankle Foundation (AOFAS) will also be used to evaluate foot function. In this scale, which is a 100-point scoring system that evaluates pain, function, and alignment, 90-100 points are excellent, 75-89 points are good, 50-74 points are good, and less than 50 points indicate poor status.
Change in lower extremity functional level | change from baseline Lower extremity functional level at 6 weeks
  The Lower Extremity Functionality Scale (LEFS), which is used in individuals with lower extremity problems, will be used to classify the functional status of individuals. AEFS is a 5-point Likert scale consisting of 20 questions. High scores in this scale, which has been adapted to Turkish and whose scoring ranges from 0 to 80, represent a better functional situation
Change in gait parameters | change from baseline temporo-spatial gait parameters at 6 weeks
  Individuals' gait will be assessed using the GAITRite® computerized walking path (CIR System INC. Clifton, NJ 07012). Data from the system, which has 18,432 sensors, is obtained by pressure-activated sensors at a rate of 60-120 Hz. In order to eliminate the learning effect, the subjects will be asked to walk at the pace they choose after three attempts are made. Rest breaks will be given between assessments and the average of three repetitions of the walk will be recorded
Change in balance | change from baseline postural sway and limits of stability at 6 weeks
  Stability limits of individuals will be evaluated with Bertec Balance Check Trainer. Participants will be asked to lie on this device in the front, back, right and left directions as far as they can go without losing their balance and without lifting the soles of their feet off the platform, and the measurement results will be recorded by the system. Also, Postural sway of individuals will be evaluated and recorded with the Bertec Balance Check Trainer. It will be evaluated in four different conditions: flat ground with eyes open, flat ground with eyes closed, soft ground with eyes open and soft ground with eyes closed. Individuals will be asked to stand upright for 10 seconds for each situation, and the results will be recorded in centimeters by the system (Force plate AM, Bertec, Columbus, OH).

CONTACTS AND LOCATIONS:
Overall Officials: Gul Yazicioglu, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No